CLINICAL TRIAL: NCT05653141
Title: Prediction of Post-stroke Cognitive Decline and Dementia: Impact of Cognitive Reserve and Post-stroke Life Style
Brief Title: Post-stroke Cognitive Impairment
Acronym: CogStroke
Status: Active, not recruiting | Type: Observational
Sponsor: Roza Umarova (Other)
Responsible Party: Sponsor-Investigator, Roza Umarova, PD Dr., Principal Investigator, Head of out-patient clinic of cognitive neurology, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: Studien-Nr. 4599
Record Dates: First submitted 2022-11-23; First posted 2022-12-16 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: First-ever Ischemic Stroke; Cognitive Performance
Keywords: Ischemic stroke; Cognitive reserve
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke patients: Adults with first-ever anterior circulation stroke

SUMMARY:
Present study aims to track the post-stroke cognitive trajectories and to investigate its inter-individual variability.

DETAILED DESCRIPTION:
The study aim is to establish a model capturing patients' inter-individual variability in susceptibility to stroke damage to predict stroke-induced cognitive trajectories. This is a prospective longitudinal observational national monocentric study for 6 years (recruitment during the first 3 years). The investigators perform comprehensive neuropsychological testing in i) acute stroke phase (0-10 days post-stroke), ii) sub-acute stroke phase (3 months post-stroke), and iii) chronic stroke phase (12 months and 3 years post-stroke). At each time point, cognitive performances as well as clinical and functional status will be assessed. Furthermore, the investigators will assess the proxies of cognitive reserve and the level of post-stroke physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* First-ever anterior circulation ischemic stroke confirmed by routine MRI
* Time of enrollment: ≤ 10 days from stroke onset.

Exclusion Criteria:

* Previous stroke anamnestic or based on clinical imaging
* Additional stroke in posterior circulation
* Conditions that preclude the cognitive testing (e.g. delirium, intubation, reduced vigilance
* Neurological or psychiatric conditions that preclude the data interpretation (e.g. pre-stroke dementia, schizophrenia, brain tumor, regular intake of benzodiazepine, depression)
* MRI contraindication
* Native language other than German, French or Italian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study recuits patients hospitalized at the Department of Neurology of the University Hospital of Bern (Inselspital)
Sampling Method: Non-Probability Sample
Enrollment: 335 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed cognitive deterioration (DCD) | at 3 months, at 12 months and at 36 months post-stroke
  The investigators will assess number of participants with deterioration of the cognitive performance in ≥2 cognitive domains on ≥ 1 Standard Deviation (1 SD).
Number of participants with delayed functional deterioration | at 3 months, at 12 months and at 36 months post-stroke
  The investigators will assess number of participants with deterioration of functional disability will be defined as decrease in disability level to one point assessed via modified Rankin Scale (mRS, 0-6, whereas 0=no functional disability).

SECONDARY OUTCOMES:
Number of participants with post-stroke cognitive impairment | 10 days post-stroke, 3 months, 12 months and at 36 months post-stroke
  The investigators will assess number of participants with post-stroke cognitive impairment that is defined as at least moderate deficit (performance below -1.5 SD) in ≥ 2 cognitive domains. The cognitive performance across all basic cognitive domains is assessed using a standardized neuropsychological test battery with available normative data. The test battery includes tests from Consortium to Establish a Registry for Alzheimer's Disease (CERAD), Trail Making Test A + B, verbal fluency, alertness test, digit span (forward and backward), Bells test, and Montreal Cognitive Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Roza M. Umarova, PD Dr., Principal Investigator — Department of Neurology, Inselspital, University Hospital Bern, University of Bern
Locations (1):
- Department of Neurology, Inselspital, University Hospital Bern, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Umarova RM. Adapting the concepts of brain and cognitive reserve to post-stroke cognitive deficits: Implications for understanding neglect. Cortex. 2017 Dec;97:327-338. doi: 10.1016/j.cortex.2016.12.006. Epub 2016 Dec 16. PMID 28049565
- [Derived] Gallucci L, Sperber C, Monsch AU, Kloppel S, Arnold M, Umarova RM. Improving diagnostic accuracy of the Montreal Cognitive Assessment to identify post-stroke cognitive impairment. Sci Rep. 2024 Aug 29;14(1):20125. doi: 10.1038/s41598-024-71184-x. PMID 39209968